CLINICAL TRIAL: NCT07006220
Title: COPE-Spain: Project COPE (Coping Options for Parent Empowerment) Adapted for Parents With Adolescent Children in Spain
Brief Title: Project COPE-Spain (Coping Options for Parent Empowerment)
Acronym: COPE-ES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Educación a Distancia (Other)
Collaborators: IES Isaac Newton (Unknown)
Responsible Party: Principal Investigator, Julia García Escalera, Associate Professor, Universidad Nacional de Educación a Distancia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: COPE-ES
Record Dates: First submitted 2025-03-20; First posted 2025-06-05 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Anxiety Symptoms; Depressive Symptoms; Parental Stress
Keywords: adolescents; transdiagnostic; school; COPE; UP-A; UP; Unified Protocol; Spain
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COPE Group (Experimental): Participants in this group will receive the COPE (Coping Options for Parent Empowerment) Program adapted as a universal prevention program for caregivers of adolescents. The program will consist of four in-person group sessions (90 minutes each) conducted over four consecutive weeks. The program focuses on improving parents' emotional regulation, enhancing parenting skills, and fostering a positive family environment.
  Assessments will be conducted at baseline (pre-intervention), post-intervention, and at 1-month follow-up.
  Interventions: Behavioral: COPE Program
- No Intervention: Waitlist Control Group (No Intervention): Participants in this group will serve as a waitlist control and will not receive the intervention immediately. Instead, they will begin the program after the experimental group has completed it, resulting in a 4-week waiting period. During this time, they will complete an additional assessment at the 4-week mark prior to their baseline, aligning with the pre-intervention timing of the experimental group. In total, they will complete assessments at four time points: 4 weeks prior to baseline, at baseline, post-intervention, and at 1-month follow-up. After the waiting period, they will receive the same COPE program intervention, following the identical structure and session format as the experimental group.

INTERVENTIONS:
Behavioral: COPE Program — The COPE Program (Coping Options for Parent Empowerment) is a brief, structured, transdiagnostic intervention designed to enhance parents' emotional regulation skills, improve parenting strategies, and foster a positive family environment. The program consists of four in-person group sessions, each lasting 90 minutes, conducted over four consecutive weeks.
  Each session focuses on specific emotional regulation and parenting skills:
  Session 1: Understanding emotional responses and parenting strategies based on positive reinforcement, selective attention, and empathy.
  Session 2: Identifying family values, promoting healthy routines, and planning alternative parenting behaviors.
  Session 3: Practicing mindfulness techniques and modeling emotional regulation in the presence of children.
  Session 4: Addressing intolerance to uncertainty, cognitive distortions, and promoting healthy independence in adolescents.
  Arms: COPE Group

SUMMARY:
The goal of this study trial is to establish the preliminary clinical utility of the COPE program (Coping Options for Parent Empowerment) adapted for caregivers of adolescents in the Spanish context. This program aims to improve parents' emotional well-being, enhance their parenting skills, and promote positive changes in their childrens' emotional and behavioral well-being. This study will adapt the COPE program for in-person group administration in the Spanish context, specifically in the school setting.

DETAILED DESCRIPTION:
The research project, titled "COPE-Spain: Adapting Project COPE (Coping Options for Parent Empowerment) for Caregivers of Adolescents in the Spanish Context," aims to evaluate the preliminary clinical utility of Project COPE (Coping Options for Parent Empowerment). Project COPE was developed at the University of Miami, with Dr. Jill Ehrenreich-May as the Principal Investigator, and has been evaluated in several studies. This protocol consists of a brief, structured intervention delivered in four group sessions, designed to improve parents' emotional well-being, strengthen their emotional regulation skills, and foster a positive family environment. Initially, Project COPE was developed to help caregivers of children during the COVID-19 pandemic and was later administered to caregivers of children with Autism Spectrum Disorder (ASD). The present study seeks to adapt Project COPE to be administered to caregivers of adolescents (instead of children) as an in-person group program implemented in the school setting.

ELIGIBILITY:
Inclusion Criteria:

* Being a parent or legal guardian of an adolescent enrolled at IES Isaac Newton during the 2024-2025 academic year.
* Participants must have availability to attend all four program sessions at the scheduled time.

Exclusion Criteria:

* Current Psychological Treatment: the parent or legal guardian is currently receiving individual psychological treatment and/or family therapy.
* Psychiatric medication changes within 4 weeks prior to the study and/or psychiatric medication changes during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Measure of Anxiety as assessed by the OASIS | Baseline, Week 4 and up to 1 month after the program.
  The Overall Anxiety Severity and Impairment Scale is a 5 self-reported questionnaire evaluating the severity and functional impairment due to anxiety. The total score ranges from 0 (no anxiety) to 20 (severe anxiety).
Measure of Depression as assessed by the ODSIS | Baseline, Week 4 and up to 1 month after the program.
  Overall Depression Severity and Impairment Scale is a 5-item measure assessing the frequency and intensity of depressive symptoms. The total score ranges from 0-20 with the higher score indicating increased depression.
Parental Stress Scale (PSS) | Baseline, Week 4 and up to 1 month after the program.
  The Parental Stress Scale is an 18-item measure assessing parents' feelings about their parenting role, exploring both positive (e.g., emotional benefits, personal development) and negative (e.g., demands on resources, feelings of stress) aspects on parenthood. All items are rated on 5-point Likert scale from 1 (Strongly disagree) to 5 (Strongly agree). Items are summed with higher scores indicating higher levels of parental stress.
Change in parenting beliefs as measured by the PSOC Scale | Baseline, Week 4 and up to 1 month after the program.
  Parenting Sense of Competence scale is a 17-item measure of parenting self-efficacyand satisfaction. It has a total score ranging from 17 to 102 with the higher scores indicating greater self-efficacy and satisfaction in the parenting role.

SECONDARY OUTCOMES:
Parent-report of the Revised Children's Anxiety and Depression Scale (RCADS-30) | Baseline, Week 4 and up to 1 month after the program.
  The Revised Child Anxiety and Depression Scale - Parent Version (RCADS-P). The RCADS-30-Parent version is designed to assess symptoms of anxiety and depression in children and adolescents, based on parental reports. It is an adaptation of the self-reported RCADS-30 and evaluates six anxiety and mood-related dimensions: Generalized Anxiety Disorder (GAD), Panic Disorder (PD), Social Phobia (SP), Separation Anxiety Disorder (SAD), Obsessive-Compulsive Disorder (OCD), Major Depressive Disorder (MDD). The RCADS-P consists of 30 items. Each item is rated on a 4-point Likert scale ranging from 0 (never) to 3 (always), reflecting the frequency of the child's symptoms as perceived by the parent or caregiver.

OTHER OUTCOMES:
Socio-Demographic Information Questionnaire | Baseline.
End of Program Questionnaire | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Julia Garcia-Escalera, Associate Professor, Study Director — Universidad Nacional de Educación a Distancia
Locations (1):
- IES Isaac Newton, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Halliday ER, Cepeda SL, Grassie HL, Jensen-Doss A, Ehrenreich-May J. Initial Effects of a Brief Transdiagnostic Intervention on Parent Emotion Management During COVID-19. Child Psychiatry Hum Dev. 2024 Apr;55(2):372-383. doi: 10.1007/s10578-022-01409-5. Epub 2022 Aug 17. PMID 35976544
- [Background] Ehrenreich-May J, Halliday ER, Karlovich AR, Gruen RL, Pino AC, Tonarely NA. Brief Transdiagnostic Intervention for Parents With Emotional Disorder Symptoms During the COVID-19 Pandemic: A Case Example. Cogn Behav Pract. 2021 Nov;28(4):690-700. doi: 10.1016/j.cbpra.2021.01.002. Epub 2021 Feb 20. PMID 34629841